CLINICAL TRIAL: NCT03649685
Title: A Randomized Clinical Trial of Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment for Obsessive-Compulsive Disorder
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Obsessive Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: RenJi Hospital (Other); Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhen Wang, vice-president, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMHC-OCD-003
Record Dates: First submitted 2018-08-23; First posted 2018-08-28 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-04

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group1: rTMS(bilateral SMA) (Active Comparator): Continuous theta burst stimulation (cTBS) stimulation will be applied over the bilateral SMA once a day, 5 days/week, for 4 weeks.
  Interventions: Device: Continuous theta burst stimulation (cTBS)
- Group2: rTMS(right DLPFC) (Experimental): Continuous theta burst stimulation (cTBS) stimulation will be applied over the right DLPFC once a day, 5 days/week, for 4 weeks.
  Interventions: Device: Continuous theta burst stimulation (cTBS)
- Group3: rTMS(right DLPFC+bilateral SMA) (Experimental): Continuous theta burst stimulation (cTBS) stimulation will be applied over the right DLPFC and bilateral SMA once a day, 5 days/week, for 4 weeks.
  Interventions: Device: Continuous theta burst stimulation (cTBS)
- Group4: shame rTMS (Sham Comparator): The sham rTMS will be applied over the bilateral SMA once a day, 5 days/week, for 4 weeks.
  Interventions: Device: shame rTMS

INTERVENTIONS:
Device: Continuous theta burst stimulation (cTBS) — 50Hz of 90% MT for 3 pulses train over will be repeated at 200ms for the 40s, 600 pulses
  Arms: Group1: rTMS(bilateral SMA); Group2: rTMS(right DLPFC); Group3: rTMS(right DLPFC+bilateral SMA)
Device: shame rTMS — The sham coil has been specifically developed to mimic the real one but is not associated with a stimulus sensation compared to the coil delivering real stimulation cTBS.
  Arms: Group4: shame rTMS

SUMMARY:
This study will evaluate the possible therapeutic effects of repetitive transcranial magnetic stimulation(rTMS) in obsessive-compulsive disorder (OCD) in OCD patients who have not fully responded to pharmacotherapy, and the underlying neural mechanism by EEG.

DETAILED DESCRIPTION:
The purpose of study is to examine the efficacy of rTMS over different brain areas, including the bilateral supplement motor Area (SMA), the right dorsal lateral prefrontal cortex (DLPFC) and SMA+DLPFC in the treatment of OCD. 120 OCD patients will be randomized into four groups. Continuous theta burst stimulation (cTBS) stimulation will be performed once a day, five times a week, for four weeks. The investigators will assess improvement after four weeks of cTBS. Though the study, Yale-Brown Obsessive Compulsive Scale（Y-BOCS）, the Dimensional Yale-Brown Obsessive-Compulsive Scale (DY-BOCS), the Barratt Impulsiveness Scale-11 (BIS-11), the Beck Depression Inventory(BDI), the Beck Anxiety Inventory (BAI), Perceived Stress Scale(PSS), Pittsburgh sleep quality index(PSQI), the Obsessive-Compulsive Inventory-Revised(OCI-R) and side effects will be obtained by a trained investigator. The patients will also receive magnetic resonance imaging scan and electroencephalography (EEG).

ELIGIBILITY:
Inclusion Criteria:

* age>18 years old;
* DSM-5 criteria for OCD;
* Y-BOCS total score > or = 16, despite treatment with an adequate trial of a serotonin reuptake inhibitor (SRI) and currently using adequate, stable dose of SRI at least 4 weeks. An adequate SRI trial is defined as treatment for at least 12 weeks on the SRI, that meets or exceeds the recommended dosage level for OCD;
* >or＝9 yrs education

Exclusion Criteria:

* any additional current psychiatric comorbidity, except for obsessive-compulsive personality disorder
* serious suicide risk;
* the inability to receive rTMS because of metallic implants, or history of seizures，or history of head injury, or history of neurosurgery;
* any major medical disease;
* pregnancy or nursing of an infant;
* participation in current clinical study;
* current use of any investigational drug;
* TMS/DBS treatment at any point in their lifetime;
* history of long-time use of benzodiazepines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Symptom improvement assessed by the Yale-Brown Obsessive Compulsive Scale | Up to 6 months
  The responder on Y-BOCS is defined as a Y-BOCS decrease at least 25% from the baseline at post-treatment

SECONDARY OUTCOMES:
The Dimensional Yale-Brown Obsessive-Compulsive Scale (DY-BOCS) | Up to 6 months
  The DY-BOCS self-report is composed of an 88-item self-report checklist, designed to provide a detailed description of obsessions and compulsions that are divided into six different OC symptom dimensions.
The Barratt Impulsiveness Scale-11 (BIS-11) | Up to 6 months
  It is is an important tool for measuring impulsivity.
The Beck Depression Inventory(BDI) | Up to 6 months
  It is a 21-item self-report measure scored on a 4-point Likert-type scale to summarize recent symptoms of depression.
The Beck Anxiety Inventory (BAI) | Up to 6 months
  It is a 21-item self-report inventory that is used for measuring the severity of anxiety.
State-trait Anxiety Inventory(STAI) | Up to 6 months
  It has 20 items for assessing trait anxiety and 20 for state anxiety.
Perceived Stress Scale(PSS) | Up to 6 months
  It is to measure the degree to which situations in one's life are appraised as stressful.
Pittsburgh sleep quality index(PSQI) | Up to 6 months
  It is a self-report questionnaire that assesses sleep quality over a 1-month time interval.
The Obsessive-Compulsive Inventory-Revised(OCI-R) | Up to 6 months
  It's a self-report designed to measure the principal dimensions which characterise obsessive-compulsive disorder.
side effects | Up to 6 months
  It measures side effects including dizziness, headache, itching and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, PhD,MD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China